CLINICAL TRIAL: NCT04558788
Title: Analysis of Cellular Stress Markers in the Intestine of Patients With Graft-versus-host Disease
Brief Title: Cellular Stress Reactions During Graft-versus-host Disease
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director of the Division of Tumor Immunology, University of Freiburg
Other Study IDs: Cellular stress in GVHD
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Graft Vs Host Disease; Graft Versus Host Disease
Keywords: GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Uninflamed intestine: Patients who underwent diagnostic endoscopy and received a diagnosis of no intestinal inflammation
  Interventions: Diagnostic Test: Immunohistochemistry on intestinal biopsies
- Colitis: Patients with active colitis
  Interventions: Diagnostic Test: Immunohistochemistry on intestinal biopsies
- Acute GVHD: Patients with acute gastrointestinal (GI) GVHD
  Interventions: Diagnostic Test: Immunohistochemistry on intestinal biopsies

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry on intestinal biopsies — Immunohistochemistry will be performed on human intestinal biopsies

SUMMARY:
This study has the aim to analyze intestinal expression of cellular stress molecules in patients with intestinal GVHD. Patients with colitis and patients without intestinal inflammation will serve as controls.

DETAILED DESCRIPTION:
Acute graft-versus-host disease (GVHD) is a major cause of morbidity and mortality in patients undergoing allogeneic hematopoietic cell transplantation (allo-HCT). Acute GVHD results from a complex multi-step crosstalk between extensive epithelial tissue damage in the patient and activation of the allo-reactive immune system transferred with the donor graft. The conditioning treatment prior to allo-HCT creates an inflamed microenvironment with high concentrations of pathogen-associated and danger-associated molecular patterns (PAMPs and DAMPs) as well as pro-inflammatory cytokines. This inflammation is perpetuated by activation of myeloid immune cells and recruitment of allo-reactive T cells to the intestine. Enterocytes are subjected to cellular stress and undergo apoptosis. As a result, patients can develop high-voluminous diarrhea, dehydration, intestinal bleeding, hypalbuminemia, and generalized infections.

In this study, the investigators aim to analyze the expression of molecules related to different types of cellular stress in the intestine of patients with acute GVHD. The hypothesis is that some stress-related markers would be upregulated during GVHD. The results will be valuable to study the role of cellular stress reactions during acute GVHD pathogenesis or as potential biomarkers for disease activity.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years intestinal biopsy depending on cohort: healthy intestinal tissue, colitis or GVHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will recruit adults at least 18 years of age, who underwent intestinal biopsy and either had (i) non-inflamed intestinal tissue, (ii) colitis, (iii) graft-versus-host disease.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Immunohistochemical staining | 1 year
  Immunohistochemical staining

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No